CLINICAL TRIAL: NCT05312359
Title: Brain Mechanism and Intervention of Executive-control Dysfunction Caused by Impaired Prefrontal-ventral Striatum Synchronization Among Substance Dependents
Brief Title: Brain Mechanism and Intervention of Executive-control Dysfunction Among Substance Dependents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDu-010
Record Dates: First submitted 2022-03-05; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-01

CONDITIONS: Substance Dependence; Executive Function Disorder; Transcranial Alternating Current Stimulation
Keywords: Substance dependence; Execution-control dysfunction; Synchronization; Transcranial alternating current stimulation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy control group (No Intervention): No intervention is conducted in the healthy control group.
- Intervention group of amphetamine addiction (Experimental): A 20-minute tACS intervention of real-stimulus is conducted twice a day for a total of 10 days in the intervention group of amphetamine addiction.
  Interventions: Device: Transcranial alternating current stimulation-true stimulus
- Control group of amphetamine addiction (Sham Comparator): A 20-minute tACS intervention of sham-stimulus is conducted twice a day for a total of 10 days in the control group of amphetamine addiction.
  Interventions: Device: Transcranial alternating current stimulation-sham stimulus
- Intervention group of alcohol addiction (Experimental): A 20-minute tACS intervention of real-stimulus is conducted twice a day for a total of 10 days in the intervention group of alcohol addiction.
  Interventions: Device: Transcranial alternating current stimulation-true stimulus
- Control group of alcohol addiction (Sham Comparator): A 20-minute tACS intervention of sham-stimulus is conducted twice a day for a total of 10 days in the control group of alcohol addiction.
  Interventions: Device: Transcranial alternating current stimulation-sham stimulus

INTERVENTIONS:
Device: Transcranial alternating current stimulation-true stimulus — The adhesive electrodes were placed at F3 and F4 positions of the 64-bit EEG caps of the 10-20 system, corresponding to bilateral prefrontal lobes respectively. Before the intervention, the individual alpha frequency (IAF) of the subjects was measured according to the average peak value of α waves at dorsolateral prefrontal cortex in the closed state. Then an alternating current at θ frequency (θ = IAF - 5Hz) was applied to each subject based on its IAF value. The amplitude of stimulation was increased with a step of 20μA starting from 0. When the subjects had a slight prickling sensation or optical illusion, the stimulation current was decreased with a step of 20μA until the sensation disappeared. The current value at this time was used as the stimulation current of the subjects.
  Arms: Intervention group of alcohol addiction; Intervention group of amphetamine addiction
Device: Transcranial alternating current stimulation-sham stimulus — The adhesive electrodes were placed at F3 and F4 positions of the 64-bit EEG caps of the 10-20 system, corresponding to bilateral prefrontal lobes respectively. The actual stimulation waveform was just implemented in the first 60 s (or more longer) and then faded out.
  Arms: Control group of alcohol addiction; Control group of amphetamine addiction

SUMMARY:
The investigators assume that tACS could improve amphetamine and alcohol dependent patients' executive-control function by adjusting the synchronization patterns and enhancing the functional connectivity of the prefrontal-ventral striatum pathway. A random controlled trial will be used to test the effect of θ-tACS treatment. Three months follow-up assessment will be conducted to test the changing of executive-control function and its mechanism.

DETAILED DESCRIPTION:
Substance abuse has become a major social and public health problem in China, especially for amphetamine abuse and alcohol abuse. Executive-control dysfunction is the main symptom for substance dependents. Previous studies have demonstrated the relationship between cognitive dysfunction and prefrontal-ventral striatum pathway. Studies have shown that abnormal phase synchronization and phase-amplitude coupling (PAC) induced the impairment of cognitive, and tACS could improve executive-control function by adjusting the abnormal synchronization. But it has not been verified among MA or alcohol patients. The investigators assume that tACS could improve MA and alcohol dependent patients' executive-control function by adjusting the synchronization patterns and enhancing the functional connectivity of the prefrontal-ventral striatum pathway. A random controlled trial will be used to test the effect of θ-tACS treatment. Three months follow-up assessment will be conducted to test the changing of executive-control function and its mechanism. This study will provide a practical and theoretical basis for developing a novel treatment for substance dependents.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60, male or female, with 9 or more years of education, and able to complete questionnaire evaluation and behavioral tests
* Meet DSM-5 diagnostic criteria for amphetamine-type substance addiction or alcohol addiction
* Have used amphetamine or alcohol for at least one year (at least once a week)
* Normal vision and hearing, or within the normal range after correction
* Agree to cooperate in the follow-up evaluation
* No metal implantation in the head, no history of nerve problems or head injury, and no skin sensitivity

Exclusion Criteria:

* Have severe cognitive impairment, such as a history of head trauma, cerebrovascular disease, epilepsy, etc.
* Have used drugs promoting cognitive function in the last 6 months
* Have impaired intelligence (IQ<70)
* Abuse or dependence of other psychoactive substances (except nicotine) in the last 5 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of inhibitory control ability | baseline, immediately after the intervention, one month after the intervention, three months after the intervention
  The change of inhibitory control ability will be reflected by participants' performance in the Go/No Go task.
The change of theta(θ) phase synchronicity | baseline, immediately after the intervention, one month after the intervention, three months after the intervention
  The change of θ phase synchronicity in the prefrontal - ventral striatum pathway in amphetamine addicts and alcohol addicts will be measured by EEG.
The change of theta-gamma phase amplitude coupling(θ-γ PAC) | baseline, immediately after the intervention, one month after the intervention, three months after the intervention
  The change of θ-γ PAC in the prefrontal - ventral striatum pathway in amphetamine addicts and alcohol addicts will be measured by EEG.

SECONDARY OUTCOMES:
The change of working memory | baseline, immediately after the intervention, one month after the intervention, three months after the intervention
  The change of working memory will be measured by the two-back task.
DA metabolic rate | baseline
  DA metabolism was measured by Positron Emission Computed Tomography
The change of decision-making ability | baseline, immediately after the intervention, one month after the intervention, three months after the intervention
  The change of decision-making ability will be measured by the Balloon Analog Risk Task.

OTHER OUTCOMES:
The The change of depression | baseline, immediately after the intervention, one month after the intervention, three months after the intervention
  Depression will be measured by the Patient Health Questionnaire-9(PHQ-9). The total score of PHQ-9 ranged from 0 to 27, in which higher scores mean a higher level of depression.
The change of anxiety | baseline, immediately after the intervention, one month after the intervention, three months after the intervention
  Anxiety will be measured by the questionnaire of Generalized Anxiety Disorder(GAD-7). The total score of GAD-7 ranged from 0 to 21, in which higher scores mean a higher level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China